CLINICAL TRIAL: NCT03240627
Title: Double-blind, Vehicle-controlled, Randomised, Multi-centre Study to Evaluate the Efficacy and Safety of LH-8 Cutaneous Solution in Children and Adolescents With Moderate to Severe Scalp Alopecia Areata.
Brief Title: Efficacy and Safety of LH-8 in Paediatric Alopecia Areata
Acronym: AA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Legacy Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAAINBOW
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: Alopecia Areata; Pediatric Disorder
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, vehicle-controlled multicentre trial in parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LH-8 cutaneous solution (Experimental): LH-8 cutaneous solution (0.126 mL per spray) applied to the whole scalp:
  Interventions: Drug: LH-8
- Placebo cutaneous solution (Placebo Comparator): Placebo cutaneous solution (0.126 mL per spray) applied to the whole scalp:
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LH-8 — LH-8 cutaneous solution
  Arms: LH-8 cutaneous solution
Drug: Placebo — Placebo cutaneous solution
  Arms: Placebo cutaneous solution

SUMMARY:
Double-blind, randomised, multi-centre study to evaluate the efficacy and safety of LH-8 cutaneous solution versus placebo in children and adolescents with moderate to severe scalp alopecia areata.

Phase 2/3 study performed in France, Germany, Bulgaria and India in 100 patients.

DETAILED DESCRIPTION:
Methods / trial design:

Randomised, double-blind, vehicle-controlled multicentre trial in parallel groups.

At screening (Visit 0), subjects will discontinue their previous treatment for alopecia areata, if any. Screening period will last up to 28 days. The 24-week treatment phase will include assessment Visits 1 to 3, which will take place at 12-week intervals. At assessment Visit 1, eligible subjects will be randomly assigned in a 2:1 ratio to receive LH-8 cutaneous solution or vehicle (placebo) twice daily for a 24 week treatment period. During the treatment phase the subjects will complete daily their drug diaries. The post-treatment safety and efficacy follow-up phase will include Visit 4 and Visit 5, 12 and 24 weeks after end of treatment, respectively.

Subjects (as applicable) and parents will be instructed to contact the investigator, if an event on scalp (intolerance) occurs during the treatment or post-treatment period. They may be asked to come to the site for an unscheduled visit, in order to perform additional examinations.

ELIGIBILITY:
Male and female children and adolescents aged 2 to less than 18 years with active alopecia areata involving 25% to 95% of the scalp between 6 months and 3 years in duration.

Diagnosis and main criteria for inclusion: Male and female children and adolescents aged 2 to less than 18 years with active alopecia areata involving 25% to 95% of the scalp between 6 months and 3 years in duration.

Inclusion criteria:

1. Male and female children and adolescents aged 2 to less than 18 years.
2. Active scalp alopecia areata, involving 25% to 95% of the scalp (as measured by SALT score at screening).
3. Duration of hair loss between 6 months and 3 years.
4. Female subjects of childbearing potential (postmenarcheal) must have a negative urine pregnancy test at screening. Females of childbearing potential must either not be sexually active or be using an adequate birth control method throughout the duration of the study.
5. All subjects taking thyroid medication or hormonal therapy must be on a stable dose for 6 months and maintain such throughout the study.
6. Subjects must be willing to maintain the same hair style, including hair dye, throughout the study period.
7. Written informed consent signed by parent(s) or legally authorized representative and assent or consent signed by the subjects, if applicable, according to national regulations prior to any protocol specific procedures.

Exclusion criteria:

1. Hypersensitivity or intolerance to any active IMP substances (onion, citrus, caffeine, theobromine) or excipients (glycerine, betaine or ethanol).
2. Any cause of hair loss other than alopecia areata.
3. Active scalp inflammation except alopecia areata.
4. Nevi, cutaneous or non-cutaneous lesions currently undiagnosed but suspicious for malignancy.
5. Female adolescents who are pregnant or who are nursing or plan pregnancy during the trial period.
6. Use of topical medication (listed in protocol Section 10.7.1) within 2 weeks prior to Visit 1.
7. Use of systemic alopecia areata therapies (e.g. prednisone, cyclosporine, methotrexate), including use of these medications for other indications, and intralesional corticosteroids within 1 month prior to Visit 1.
8. Administration of hydroxychloroquine or finasteride within two months prior to Visit 1.
9. Use of phototherapy, laser therapy or excimer laser therapy on the scalp within three months prior to Visit 1.
10. Use of infliximab within two months, adalimumab within three months, and ustekinumab within four months prior to Visit 1 or use of other TNF inhibitors and biologic agents within one month or five half-lives before Visit 1, whichever is longer.
11. Prior treatment with IMP.
12. Evidence or history of alcohol, medication or drug abuse.
13. History of systemic or cutaneous medical, or psychiatric disease which will put subject at risk or interfere with assessments.
14. Participation in any other clinical trial within 30 days prior to Visit 1.
15. Subject is in a dependent relationship (e.g. relative or family member) with the investigator's or sponsor's staff.
16. Any other condition or circumstance that, in the opinion of the investigator, could compromise the subject's ability to comply with the study protocol.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Relative change in scalp alopecia areata severity scores (SALT) from baseline value to be assessed after 24 weeks of treatment. | 24 weeks treatment
  Visual assessment and global standardised scalp photographs for SALT evaluation.

SECONDARY OUTCOMES:
Absolute change in SALT score from baseline at the end of 24 weeks' treatment period. | 24 weeks treatment
Proportion of the responders, i.e. subjects achieving at least a 40% relative reduction in SALT score from baseline at the end of 24 weeks' treatment period. | 24 weeks treatment
Adverse events | 48 weeks
General physical examination findings, including irritation of eyes and skin | 24 weeks treatment
Visual assessment and global standardised scalp photographs for SALT evaluation. | After 12 and 24 weeks treatment
  Evaluation of duration of treatment effect in responders, measured as relative SALT score changes from Visit 3 (end of treatment) after 12 weeks (Visit 4) and 24 weeks (Visit 5) of treatment-free period. (Visual assessment and global standardised scalp photographs for SALT evaluation.)
Assessment of treatment effect on hair follicles in non-alopecic areas by quantifying the number of new alopecic areas. | 24 weeks treatment
Assessment of the rate of spontaneous hair regrowth. | For 6-12 months
  Assessment of the rate of spontaneous hair regrowth in placebo treated subjects with alopecia areata active for 6-12 months compared to those with alopecia areata active for more than 12 months. (Visual assessment and global standardised scalp photographs for SALT evaluation).
• Absolute and relative change from baseline in Children's Dermatology Life Quality Index (CDLQI) scores. | 48 weeks
Change in percentage of subjects from baseline by the severity banding CDLQI scores. | 48 weeks
Percentages of subjects by EuroQol Five Dimensions Youth Questionnaire (EQ-5D-Y) dimensions and levels at Visits 1-5. | 48 weeks
Absolute and relative change of the EQ-Visual Analogue Scale (EQ-VAS) scores from baseline | 48 weeks
Evaluation of the Paediatric Alopecia Areata Patient Benefit Index (PAAPBI) scores at Visits 1 to 5. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike BLUME-PEYTAVI, Prof. Dr., Study Chair — Charité-Universitätsmedizin Berlin, Dept Dermatology, Germany; Pascal REYGAGNE, Dr., Principal Investigator — Sabouraud Center, Saint-Louis Hospital, France; Petyo Brezoev, Dr., Principal Investigator — DDC Alexandrovska-Sofia", Bulgaria; Uwe Schwichtenberg, Dr., Study Director — Hautarztpraxis, Bremen-Vegesack, Germany; Maya Milanova, Dr, Study Director — Center of Skin and venereal diseases, Sliven, Bulgaria; Mariyana Venelinova_Rusinova, Dr, Study Director — MC Doverie, Sofia, Bulgaria; Ishad Aggarwal, Dr, Principal Investigator — Health Point Hospital 21, Kolkata, India
Locations (3):
- Multicenter Clinical Trials, Sofia, Bulgaria
- Centre Sabourand - Hospital Saint-Louis, 1, Avenue Claude Vellefaux, Paris, France
- Clinical Research Center for Hair and Skin Science, Charité-Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blume-Peytavi U, Piraccini BM, Reygagne P, Guiraud J, Mukherjee B, Guichard A, Liu J, Pralong W, Harti S. Efficacy and safety of Cinainu in paediatric alopecia areata: an international, double-blind, randomized, placebo-controlled, phase II/III trial. Br J Dermatol. 2026 Jan 6;194(1):37-46. doi: 10.1093/bjd/ljaf279. PMID 40668972